CLINICAL TRIAL: NCT00920452
Title: RELIANCE QUADRIPOLAR DEFIBRILLATION LEADS (4-SITE)FIELD FOLLOWING The 4-SITE Field Following Study (4-SITE FF)
Brief Title: The 4-SITE Field Following Study (4-SITE FF)
Acronym: 4-SITE FF
Status: Completed | Type: Observational
Sponsor: Guidant Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 4-SITE FF 0209
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2010-11

CONDITIONS: ICD and CRT-D Indicated Patients
Keywords: implantable cardioverter defibrillator (ICD); defibrillation leads, cardiac resynchronization therapy (CRT)

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate and document appropriate clinical performance of the new 4-SITE Header / Lead interface in the TELIGEN 100 HE 4-SITE (VR and DR) implantable cardioverter defibrillator (ICD) PGs (Models F103; F111), the COGNIS 100 HE 4-SITE cardiac resynchronization therapy ICD (CRT-D) PG (Model P108) when connected to any of the RELIANCE Quadripolar (4-SITE) defibrillation leads.

Appropriate clinical performance of system components of the 4-SITE systems other than the new 4-SITE header / lead interface has been evaluated and documented already in the previously conducted COGNIS and TELIGEN 100 HE FIELD FOLLOWING STUDY, The COGENT-4 Field Following Study.

Data collected may be used to support international regulatory submissions including the FDA and the Japanese Ministry of Health, Labour and Welfare.

DETAILED DESCRIPTION:
The following devices will be used (all are CE-marked):

* TELIGEN 100 HE 4-SITE (Single and Dual Chamber ICD)

  * Model Number: F103 (Quadripolar, VR);
  * Model Number: F111 (Quadripolar, IS-1, DR)
* COGNIS 100 HE 4-SITE (CRT-D)

  o Model Number: P108 (Quadripolar, IS-1, IS-1)
* RELIANCE 4-SITE leads (12 different model numbers in total as shown in the table below)

ELIGIBILITY:
Inclusion Criteria:

Study Specific:

* ICD / CRT-D Indication according to normal clinical practice
* Patients receiving:
* a single or dual chamber 4-SITE compatible ICD
* or a 4-SITE compatible CRT-D
* one of the RELIANCE 4-SITE defibrillation leads
* Patients currently implanted with a pacemaker
* upgraded to a 4-SITE compatible ICD or CRT-D (4-SITE header)
* one of the RELIANCE 4-SITE defibrillation leads

General:

* Willing and capable of providing informed consent for
* undergoing a 4-SITE system implant,
* participating in all testing associated with this clinical investigation at an approved clinical investigational centre and at the intervals defined by this protocol
* Geographically stable patients who are available for follow-up at a study centre
* Age 18 or above, or of legal age to give informed consent specific to national law

Exclusion Criteria:

Study Specific:

* ICD and CRT-D Patients scheduled for a device replacement
* CRM Patients who have or who would need an lead adaptor
* All patients who have an active or non-active defibrillation lead other than 4-SITE

General:

* Not willing and not capable of providing informed consent, undergoing a device implant, participating in all testing associated with this clinical investigation (including VT/VF shock conversion) at an approved clinical investigational centre and at the intervals defined by this protocol
* Patients who were in NYHA Class IV during the last 3 month
* Patients with pre-existing diseases, which may confound study results
* Patients currently requiring dialysis,
* Cancer patients
* Patients with drug and/or alcohol abuse history
* Life expectancy < 12 months (or expected heart transplant within 12 months)
* Patients on a Heart Transplant List
* Women who are pregnant or plan to become pregnant. Method of assessment per physician discretion.
* Enrolled in any other concurrent study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study Population: Patients should be selected from the investigator's general population indicated for an ICD or CRT-D Implantation. The investigator has the responsibility of screening all potential patients and selecting those who meet study eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 430 (Actual)
Dates: Start 2009-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Appropriate Detection of induced VT | At Implant or during VT/VF testing up to one month after implant
  Induced mean VT/VF detection time < 4.5 seconds
Appropriate induced VT/VF Shock Conversion | At Implant or during testing within one month after implant
  Successful VT/VF conversions (with 41 J, no external shock) will be 93% or higher
Appropriate pacing thresholds at follow-up with the 4-SITE defibrillation leads | entire duration of the study
  Mean pacing threshold post implant ≤ 1.5V
Appropriate Lead Impedances as a measure of lead integrity over 12 month time | entire study duration
  * Shocking lead impedance should be within the range of 20 and 80 OHM
  * Pace /sense lead impedance within 200 and 2000 OHM
Appropriate sensing and absence of artefacts | entire duration of study
  Appropriate sensing and absence of artefacts during standardized pocket manipulations and standardized provocative maneuvers during FU

CONTACTS AND LOCATIONS:
Locations (1):
- Bad Oeynhausen Herz- und Diabeteszentrum Nordrhein-Westfalen, Bad Oeynhausen, North Rhine-Westphalia, Germany